CLINICAL TRIAL: NCT02680223
Title: Efficacy of Coloured Overlays and Lenses for Adults With Reading Difficulty
Brief Title: Efficacy of Coloured Overlays and Lenses for Reading Difficulty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BA_2015
Record Dates: First submitted 2016-02-02; First posted 2016-02-11 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2019-08

CONDITIONS: Vision Disorders; Reading Disabilities
MeSH Terms: conditions — Vision Disorders; Dyslexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precision tinted lenses (Active Comparator): Precision tinted lenses will be provided for one month.
  Interventions: Device: Precision tinted lenses
- Non-beneficial tinted lenses (Sham Comparator): Tinted lenses at a colour different from but not easily distinguishable from the precision tinted will be provided for one month.
  Interventions: Device: Non-beneficial tinted lenses

INTERVENTIONS:
Device: Precision tinted lenses — Tinted lens for patient with reading difficulty or visual stress
  Arms: Precision tinted lenses
Device: Non-beneficial tinted lenses — Tinted lenses that are unlikely to help reading difficulty or visual stress
  Arms: Non-beneficial tinted lenses

SUMMARY:
This is a randomised controlled trial with the aim of testing the efficacy of coloured overlays and coloured lenses for the relief of visual stress and reading difficulties in children and young adults.

DETAILED DESCRIPTION:
Participants will be adults aged from 8 years, with symptoms of visual stress (discomfort when reading or experiencing perceptual symptoms when reading such as letters moving or distorted) or with a diagnosed reading difficulty (dyslexia). Participants will be recruited from the City University London optometry clinic and the City University London Learning Success unit. Participants within this age range and with visual stress will be eligible to participate. Potential participants with an ocular or systemic condition with possible impact on vision (e.g. amblyopia or diabetes respectively) or with intellectual disability will be excluded from the study. Each potential participant will undergo an eye examination prior to participation, during which the following tests will be conducted:

Prior to study entry:

History and symptoms Direct ophthalmoscopy (to check for ocular abnormality) Retinoscopy and subjective refraction (to quantify corrected and uncorrected refractive error) Cover tests (to look for any eye misalignment)

Baseline tests on study entry:

Each eligible participant who agrees to take part in the study will undergo testing with coloured overlays, to determine whether a particular overlay appears to be beneficial in terms of reducing difficulty or discomfort while reading. If so, the participant will be provided with the overlay to use for a period of two weeks, to determine whether it is consistently beneficial when reading during that period. In addition, the Wilkins Rate of Reading Test (WRRT) will be carried out at this baseline stage with and without the overlay.

Follow-up test 1:

The participant will attend a further appointment at the two week time point, and if the overlay was beneficial, an addition test will be carried out using the Intuitive Colorimeter, to determine the exact hue, saturation and intensity of coloured lenses that offer the most relief from difficulty or discomfort while reading. Once this colour has been determined, the hue will be modified to find the closest colour at which the participant first loses benefit (the point at which the discomfort or difficulty returns). Each colour setting (beneficial and non-beneficial) will be noted and the participant will be provided with spectacle lenses tinted exactly to one of these colour specifications. In a crossover design, the order in which true or control lenses will be provided to each participant will be determined by random number generation. Allocation will be carried out by personnel who are not researchers on this study, and who know the order (true lens tint first or second) as 1 and 2. Ordering of tinted spectacles will be handled by the personnel who are not researchers on the study, and this information will not be accessible by the researchers. Thus, tinted lens ordering will not be shared with the researchers, who will not know whether each participant is wearing the beneficial or non-beneficial tint, and so will be masked. Similarly, participants will be unaware whether they are wearing the true or control tint, at any time during their participation. The non-beneficial tint will be very similar to the beneficial tint, so neither researchers nor participants will be able to determine this. On this occasion the participant will also be asked to describe the difficulties he/she has experiences when reading with and without the coloured overlay.

Follow-up test 2:

After one month wearing the first pair of tinted lenses, reading speed will be measured again with the first pair of tinted lenses, and the participant will be asked again about their experience of reading difficulties while wearing these glasses. The participant will be asked to spend one week without any tinted lenses, and to return for a further visit after that week. After this period, the second pair of tinted lenses will be provided, to be worn for a further month.

Follow-up test 3:

Reading speed will be measured again with the second pair of tinted lenses and the participant will again be asked about their experience of reading difficulties while wearing these glasses.

Statistical analysis The main outcome measures are rates of reading provided by the two reading tests, with the two tinted lens types, the overlay, and without any tint. These are quantitative tests and the results will be compared between the two groups using an unpaired t-test, and within individuals (between baseline and follow-up tests) using a repeated measures analysis of variance. In addition, qualitative data are obtained from participants' descriptions of their experience of reading difficulty at different stages of the study. These responses will be analysed using NVivo software to look for themes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with visual stress or reading disability aged 8 years and over.

Exclusion Criteria:

* Ocular or systemic disease
* Intellectual disability

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Rate of reading | 3 months
  Wilkins rate of reading test

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Suttle, Principal Investigator — City, University of London
Locations (1):
- City University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkins AJ, Evans BJ, Brown JA, Busby AE, Wingfield AE, Jeanes RJ, Bald J. Double-masked placebo-controlled trial of precision spectral filters in children who use coloured overlays. Ophthalmic Physiol Opt. 1994 Oct;14(4):365-70. PMID 7845693
- [Background] Evans BJ, Stevenson SJ. The Pattern Glare Test: a review and determination of normative values. Ophthalmic Physiol Opt. 2008 Jul;28(4):295-309. doi: 10.1111/j.1475-1313.2008.00578.x. PMID 18565084
- [Background] Bouldoukian J, Wilkins AJ, Evans BJ. Randomised controlled trial of the effect of coloured overlays on the rate of reading of people with specific learning difficulties. Ophthalmic Physiol Opt. 2002 Jan;22(1):55-60. doi: 10.1046/j.1475-1313.2002.00002.x. PMID 11829008
- [Background] Monger L, Wilkins A, Allen P. Identifying visual stress during a routine eye examination. J Optom. 2015 Apr-Jun;8(2):140-5. doi: 10.1016/j.optom.2014.10.001. Epub 2014 Nov 11. PMID 25455572
- [Background] Allen PM, Dedi S, Kumar D, Patel T, Aloo M, Wilkins AJ. Accommodation, pattern glare, and coloured overlays. Perception. 2012;41(12):1458-67. doi: 10.1068/p7390. PMID 23586285
- [Background] Wilkins AJ, Jeanes RJ, Pumfrey PD, Laskier M. Rate of Reading Test: its reliability, and its validity in the assessment of the effects of coloured overlays. Ophthalmic Physiol Opt. 1996 Nov;16(6):491-7. PMID 8944196
- [Background] Creavin AL, Lingam R, Steer C, Williams C. Ophthalmic abnormalities and reading impairment. Pediatrics. 2015 Jun;135(6):1057-65. doi: 10.1542/peds.2014-3622. PMID 26009619